CLINICAL TRIAL: NCT01447342
Title: A Study to Evaluate the Safety and Effectiveness of the Cryo-Touch II Device for the Treatment of Forehead and/or Glabellar Lines
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MS-4400
Record Dates: First submitted 2011-09-29; First posted 2011-10-06 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Facial Wrinkles; Skin Aging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Cryo-Touch II — Percutaneous treatment with the device

SUMMARY:
A prospective, non-randomized, multicenter study to evaluate the safety and effectiveness of the cryo-touch II device for the treatment of forehead and/or glabellar lines

ELIGIBILITY:
Inclusion Criteria:

1. Subject is a male or female, 30 to 70 years old.
2. Subject is willing and able to give written informed consent.
3. Subject has a forehead wrinkle rating by the investigator/designee of at least "2" in animation on the 5-point Wrinkle Scale (5WS) which upon physical manipulation/separation of the skin demonstrates a reduction in wrinkle severity. Subject may also have a glabellar score of "1" or higher in animation on a 4-point scale.
4. Subject is willing and able to comply with study instructions and commit to all follow-up visits for the duration of the study.
5. Subject is in good general health and free of any disease state or physical condition that might impair evaluation of forehead and/or glabellar wrinkle rating or which, in the investigator's opinion, exposes the subject to an unacceptable risk by study participation.

Exclusion Criteria:

1. Subject is currently enrolled in an investigational drug or device study.
2. Subject has used an investigational drug or investigational device treatment within 30 days prior to first administration of the device.
3. Subject has a clotting disorder or has used an anticoagulant (e.g., Coumadin, clopidogrel, etc.) within seven (7) days prior to administration of the device.
4. Subject has used aspirin, or non-steroidal anti-inflammatory drugs (NSAIDs, e.g., ibuprofen, and naproxen) within seven (7) days prior to administration of the device.
5. Subject has had prior surgery that alters the subcutaneous anatomy of the target treatment sites.
6. Subject has undergone another facial cosmetic procedure at or above the level of the cheekbones within the past six (6) months.
7. Subject has any of the following conditions:

   1. History of facial nerve palsy,
   2. Marked facial asymmetry,
   3. Ptosis,
   4. History of neuromuscular disorder,
   5. Chronic dry eye symptoms,
   6. Allergy or intolerance to lidocaine,
   7. Other local skin condition (e.g., skin infection) at target treatment site,
   8. Any physical or psychiatric condition that in the investigator's opinion would prevent adequate study participation.
   9. Chronic medical condition that in the investigator's opinion would affect study participation (such as diabetes, hepatitis, HIV, etc.).
   10. Any chronic condition contraindicated for the use of nerve mapping device including heart disease, use of a cardiac pacemaker, and pregnancy.
8. Subject is known to be noncompliant or is unlikely to comply with the requirements of the study protocol (e.g., due to alcoholism, drug dependency, mental incapacity) in the opinion of the investigator.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2011-09; Primary Completion 2012-01 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Effectiveness success | Up to 4 months
  Effectiveness endpoint: wrinkle severity in the forehead in animation at 30 days post-treatment (Visit 5) as rated by the investigator/designee using the 5-point Wrinkle Scale (5WS).
Safety success | Up to 4 months
  Safety endpoint: Tolerability of treatment (LSRs), local and systemic adverse events will be assessed at all visits. Incidence of serious adverse events (SAEs) and unanticipated adverse device effects (UADEs) will be recorded. A serious adverse event is one that meets the ISO definition of SAE .

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Macro, Llc, Beverly Hills, California
  - The Aesthetics Research Center, Redwood City, California
  - Roseville Facial Plastic Surgery, Roseville, California